CLINICAL TRIAL: NCT04545554
Title: An Open-label, Ascending Multiple-dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Romosozumab in Children and Adolescents With Osteogenesis Imperfecta
Brief Title: Study to Evaluate Romosozumab in Children and Adolescents With Osteogenesis Imperfecta
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20160227; 2017-004972-74 (EudraCT Number)
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-10

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — romosozumab; Calcium; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Romosozumab: 12 - < 18 Years of Age (Experimental): Participants will receive 1 of 3 dose levels of romosozumab. All participants also received calcium and vitamin D.
  Interventions: Drug: Romosozumab; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D
- Romosozumab: 5 - < 12 Years of Age (Experimental): Participants will receive 1 of 3 dose levels of romosozumab. All participants also received calcium and vitamin D.
  Interventions: Drug: Romosozumab; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Romosozumab — Participants will receive multiple doses of romosozumab via a SC injection.
Dietary Supplement: Calcium — All participants will receive daily supplements of elemental calcium.
Dietary Supplement: Vitamin D — All participants will receive daily supplementation with vitamin D.

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) profile following multiple subcutaneous (SC) doses of romosozumab in children and adolescents with Osteogenesis Imperfecta (OI).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female children 5 to less than 18 years of age upon entry into screening
* Clinical diagnosis of OI defined as a clinical history consistent with type I-IV OI as determined by presence of expected phenotype and lack of additional features unrelated to type I-IV OI

Exclusion Criteria

* History of an electrophoresis pattern inconsistent with type I to type IV OI
* History of known mutation in a gene other than collagen type I alpha 1/collagen type I alpha 2 (COL1AI/COL1A2) causing OI or other metabolic bone disease
* History of other bone diseases that affect bone metabolism (eg, osteoporosis pseudoglioma syndrome, idiopathic juvenile osteoporosis, osteopetrosis, hypophosphatasia)
* History of Kawasaki disease, rheumatic myocarditis, ischemic cardiomyopathy, inherited cardiomyopathies, nephrotic syndrome, familial hypercholesterolemia, stroke, or any thromboembolic disorder
* Unhealed fracture as defined by orthopedic opinion
* Symptoms associated with skull abnormalities such as basilar invagination, basilar impression or Chiari malformation
* Prior treatment with anti-sclerostin antibody, fluoride or strontium, parathyroid hormone (PTH) within 12 months prior to screening, denosumab within 12 months or zoledronic acid within 6 months prior to first dose
* Less than 2 evaluable vertebrae by DXA evaluation in the region of interest, L1 - L4, as confirmed by the central imaging laboratory.
* Clinically significant valvular heart disease based on local echocardiogram (ECHO) results.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- United States (3):
  - Riley Hospital for Children, Indianapolis, Indiana
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Kepler Universitaetsklinikum GmbH, Linz, Austria
- Uniklinik Köln, Cologne, Germany
- General Children Hospital Panagioti and Aglaias Kyriakou, Athens, Greece
- Semmelweis Egyetem, Budapest, Hungary
- IRCCS Ospedale Pediatrico Bambino Gesu, Roma, Italy
- Spain (4):
  - Hospital de Cruces, Barakaldo, Basque Country
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
- Turkey (Türkiye) (3):
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Koc Universitesi Hastanesi, Istanbul
  - Ege Universitesi Ilac Gelistirme ve Farmakokinetik Arastirma Uygulama Merkezi (ARGEFAR), Izmir

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Tabaie SA, O'Mara AE, Sheppard ED, Tosi LL. A Comprehensive Review of Bone Health in a Child: From Birth to Adulthood. J Am Acad Orthop Surg. 2024 May 1;32(9):363-372. doi: 10.5435/JAAOS-D-23-00853. Epub 2024 Jan 23. PMID 38261781
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 15 study centers in Austria, Germany, Greece, Hungary, Italy, Spain, Turkey, and the United States, and participated from 21 January 2021 until 30 March 2023.
Pre-assignment Details: Ambulatory children (5 to < 12 years of age) and adolescents (12 to < 18 years of age) with osteogenesis imperfecta were enrolled to receive 1 of 3 subcutaneous (SC) dose levels of romosozumab. Specific doses are blinded due to the protection of propriety information.
Groups:
- Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age); Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age): Participants received multiple SC doses of romosozumab Dose A (low dose).
- Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age); Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age): Participants received multiple SC doses of romosozumab Dose B (medium dose).
- Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age); Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age): Participants received multiple SC doses of romosozumab Dose C (high dose).
Period: Overall Study
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Started | 4 | 4 | 4 | 5 | 4 | 4
Received at Least 1 Dose Romosozumab | 4 | 4 | 4 | 5 | 4 | 4
Received All Doses of Romosozumab | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.9) | 6.0 (1.4) | 14.3 (0.5) | 8.4 (2.4) | 14.0 (1.8) | 6.5 (0.6) | 10.5 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 4 | 2 | 1 | 9
  Male | 3 | 4 | 3 | 1 | 2 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 4 | 4 | 4 | 3 | 3 | 4 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 4 | 4 | 4 | 4 | 4 | 2 | 22
  Other | 0 | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Romosozumab
Description: Mean Cmax values following Days 1 and 57 are presented.
Time Frame: Single blood samples were taken on days 1, 8, 15, 29, 57, 64, 71, 85, 113, and 169 (end of study); pre-specified PK analysis took place on Days 1 and 57
Population: Pharmacokinetic (PK) Analysis Set: all participants for whom at least 1 PK parameter or endpoint could be adequately tested.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
μg/mL
  Day 1 | 2.64 (1.06) | 1.74 (0.825) | 13.8 (6.32) | 10.3 (1.70) | 25.7 (3.02) | 21.3 (6.45)
  Day 57 | 2.43 (1.36) | 5.55 (2.11) | 12.8 (6.31) | 9.14 (7.50) | 22.8 (10.5) | 19.4 (2.14)

2. Primary Outcome: Time to Cmax (Tmax) of Romosozumab
Description: Median tmax values following Days 1 and 57 are presented.
Time Frame: as for outcome 1
Population: PK Analysis Set: all participants for whom at least 1 PK parameter or endpoint could be adequately tested.
Measure: Median (Full Range); unit: day
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
day
  Day 1 | 6.5 [5.9 to 7.9] | 7.9 [7.9 to 15] | 6.9 [6.9 to 7.0] | 6.9 [4.9 to 7.1] | 7.0 [4.9 to 8.0] | 7.5 [6.9 to 8.9]
  Day 57 | 7.0 [7.0 to 12] | 7.0 [6.9 to 7.0] | 7.0 [6.0 to 7.9] | 8.0 [6.0 to 11] | 7.0 [4.0 to 12] | 7.5 [6.0 to 8.8]

3. Primary Outcome: Area Under the Serum Concentration Time Curve (AUC) From Time 0 to Day 28 (AUC[0-28]) of Romosozumab
Description: Mean AUC(0-28) values following Days 1 and 57 are presented.
Time Frame: Single blood samples were taken on days 1, 8, 15, 29, 57, 64, 71, and 85; pre-specified PK analysis took place on Days 1 and 57
Population: PK Analysis Set: all participants for whom at least 1 PK parameter or endpoint could be adequately tested.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
day*μg/mL
  Day 1 | 30.9 (13.5) | 16.9 (5.78) | 163 (89.1) | 113 (50.3) | 344 (106) | 234 (93.7)
  Day 57 | 27.4 (15.1) | 50.5 (20.7) | 153 (86.7) | 95.1 (76.1) | 293 (134) | 203 (40.7)

4. Primary Outcome: Accumulation Ratio of Romosozumab
Description: The accumulation ratio was calculated as AUC(0-28) at Day 57/AUC(0-28) at Day 1. Mean accumulation ratio values based on analysis at Days 1 and 57 are presented, as pre-specified.
Time Frame: as for outcome 3
Population: PK Analysis Set: all participants for whom at least 1 PK parameter or endpoint could be adequately tested.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
ratio | 0.885 (0.487) | 3.6 (2.56) | 0.922 (0.0673) | 0.724 (0.392) | 0.843 (0.260) | 0.935 (0.283)

5. Primary Outcome: Terminal Half-life of Romosozumab
Description: Median terminal half-life values at Day 57 are presented.
Time Frame: Single blood samples were taken on days 1, 8, 15, 29, 57, 64, 71, 85, 113, and 169 (end of study); pre-specified PK analysis took place on Day 57
Population: PK Analysis Set: all participants for whom at least 1 PK parameter or endpoint could be adequately tested. Data is presented for participants with evaluable data.
Measure: Median (Full Range); unit: day
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 0 | 2 | 0 | 1 | 3 | 0
day |  | 9.41 [7.62 to 11.2] |  | 7.01 [7.01 to 7.01] | 6.11 [5.58 to 6.56] |

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were adverse events (AEs) that started on or after first dose of investigational product up to the end of study (up to Day 169). Any clinically significant changes in vital signs, electrocardiogram parameters, physical exam findings, and clinical laboratory parameters were reported as TEAEs.
  Injection site reactions were events of interest (EOI) for this study.
Time Frame: Day 1 to end of study (up to Day 169); median duration on study was 5.55 months
Population: Safety Analysis Set: all participants enrolled in the study who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
Participants
  Any TEAE | 1 | 1 | 2 | 4 | 1 | 3
  Any Treatment-emergent EOI | 0 | 0 | 0 | 0 | 1 | 1

7. Secondary Outcome: Number of Participants With Changes From Baseline in Cranial Nerve VII Examination Findings at Day 57, Day 85, and Day 169
Description: Facial nerve (cranial nerve VII) function was assessed clinically by facial symmetry inspection at rest, followed by assessment of the symmetry of specific facial movements: raising eyebrows, closing the eyes, blowing out the cheeks, smiling, pursing and closing the lips. Results of the cranial nerve examination were classed as 0 = Normal; 1 = Abnormal not clinically significant; and 2 = Abnormal clinically significant. An increase from baseline indicates an increase in abnormal clinical findings on the cranial nerve VII examination.
Time Frame: Baseline (Day 1), Day 57, Day 85, and Day 169
Population: Safety Analysis Set: all participants enrolled in the study who received at least 1 dose of investigational product. Participants with data available at each time point are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
Participants
  Day 57: Blowing out of cheeks - No change (0) | 4 | 4 | 4 | 3 | 4 | 4
  Day 57: Blowing out of cheeks - Undetermined | 0 | 0 | 0 | 2 | 0 | 0
  Day 57: Closing eyes - No change (0) | 4 | 4 | 4 | 3 | 4 | 4
  Day 57: Closing eyes - Undetermined | 0 | 0 | 0 | 2 | 0 | 0
  Day 57: Closing of lips - No change (0) | 4 | 4 | 4 | 3 | 4 | 4
  Day 57: Closing of lips - Undetermined | 0 | 0 | 0 | 2 | 0 | 0
  Day 57: Pursing of lips - No change (0) | 4 | 4 | 4 | 3 | 4 | 4
  Day 57: Pursing of lips - Undetermined | 0 | 0 | 0 | 2 | 0 | 0
  Day 57: Raising eyebrows - No change (0) | 4 | 4 | 4 | 3 | 4 | 4
  Day 57: Raising eyebrows - Undetermined | 0 | 0 | 0 | 2 | 0 | 0
  Day 57: Smiling - No change (0) | 4 | 4 | 4 | 3 | 4 | 4
  Day 57: Smiling - Undetermined | 0 | 0 | 0 | 2 | 0 | 0
  Day 85: Blowing out of cheeks - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85: Blowing out of cheeks - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 85: Closing eyes - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85: Closing eyes - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 85: Closing of lips - No change (0) | 4 | 3 | 4 | 4 | 4 | 4
  Day 85: Closing of lips - Increase (to 1) | 0 | 1 | 0 | 0 | 0 | 0
  Day 85: Closing of lips - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 85: Pursing of lips - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85: Pursing of lips - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 85: Raising eyebrows - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85: Raising eyebrows - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 85: Smiling - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85: Smiling - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 169: Blowing out of cheeks - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169: Blowing out of cheeks - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 169: Closing eyes - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169: Closing eyes - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 169: Closing of lips - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169: Closing of lips - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 169: Pursing of lips - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169: Pursing of lips - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 169: Raising eyebrows - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169: Raising eyebrows - Undetermined | 0 | 0 | 0 | 1 | 0 | 0
  Day 169: Smiling - No change (0) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169: Smiling - Undetermined | 0 | 0 | 0 | 1 | 0 | 0

8. Secondary Outcome: Number of Participants With Anti-romosozumab Antibodies
Description: Treatment-boosted anti-romosozumab antibody was defined as binding antibody positive at baseline with a >4 x increase in magnitude post-baseline. Transient results were defined as negative results at the participant's last time point tested within the study period.
Time Frame: Blood samples for anti-romosozumab antibodies were taken Day 1, Day 15, Day 29, Day 85, and Day 169
Population: Safety Analysis Set: all participants enrolled in the study who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
Participants
  Binding antibody positive anytime | 0 | 1 | 2 | 0 | 1 | 1
  Neutralizing antibody positive anytime | 0 | 0 | 2 | 0 | 1 | 0
  Binding antibody positive at/before baseline | 0 | 0 | 0 | 0 | 0 | 0
  Neutralizing antibody positive at/before baseline | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-boosted antibody positive | 0 | 0 | 0 | 0 | 0 | 0
  Binding antibody positive post-baseline with negative/no results at baseline | 0 | 1 | 2 | 0 | 1 | 1
  Transient binding antibody positive post-baseline with negative/no results at baseline | 0 | 0 | 0 | 0 | 0 | 0
  Neutralizing antibody positive post-baseline with a negative/no result at baseline | 0 | 0 | 2 | 0 | 1 | 0
  Transient neutralizing antibody positive post-baseline with a negative/no result at baseline | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage Change From Baseline in Serum Concentrations of Serum Type 1 Collagen C-Telopeptide (CTX)
Description: Serum concentrations of the bone turnover marker CTX were determined at pre-specified time points.
Time Frame: Blood samples were taken Days 1 (baseline), 8, 15, 29, 57, 64, 71, 85, 113, and 169
Population: PD Analysis Set: all participants for whom at least 1 PD parameter or endpoint could be adequately estimated. Participants with data available at each time point are presented.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
percentage change
  Day 8: number analyzed (Participants) | 4 | 3 | 4 | 5 | 4 | 4
  Day 8 | 2.65 (27.91) | -19.93 (33.97) | 8.79 (19.21) | -19.38 (20.01) | -12.33 (12.93) | 7.14 (29.89)
  Day 15: number analyzed (Participants) | 3 | 4 | 4 | 4 | 4 | 3
  Day 15 | 12.26 (28.20) | -3.24 (41.30) | -2.14 (52.91) | -20.24 (21.12) | -17.22 (17.39) | 42.62 (54.95)
  Day 29: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 29 | -4.67 (21.35) | -6.67 (39.99) | 26.00 (15.11) | -7.43 (18.63) | -16.09 (27.05) | 3.76 (24.72)
  Day 57: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 57 | 1.03 (34.14) | -7.34 (25.32) | -0.32 (32.21) | -7.66 (13.16) | -1.40 (38.10) | 44.17 (95.30)
  Day 64: number analyzed (Participants) | 3 | 4 | 4 | 3 | 3 | 2
  Day 64 | -13.37 (36.33) | -18.26 (49.19) | 19.91 (43.95) | -10.60 (36.12) | 10.95 (23.38) | -28.14 (11.51)
  Day 71: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 4
  Day 71 | 18.20 (53.85) | -25.30 (50.43) | 35.26 (68.16) | -3.37 (8.25) | 15.14 (51.39) | 60.12 (106.28)
  Day 85: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85 | -10.56 (22.18) | -37.50 (14.12) | 9.95 (30.71) | 5.08 (24.34) | 0.71 (44.55) | 15.77 (58.40)
  Day 113: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 113 | -3.83 (22.30) | -30.38 (19.59) | 25.94 (39.76) | 6.98 (37.98) | 7.03 (40.23) | -19.58 (10.98)
  Day 169: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169 | -6.15 (54.87) | -29.78 (31.60) | -1.72 (40.42) | 11.08 (16.19) | -8.07 (16.73) | 8.08 (49.45)

10. Secondary Outcome: Percentage Change From Baseline in Serum Concentrations of Procollagen Type 1 N-terminal Propeptide (P1NP)
Description: Serum concentrations of the bone turnover marker P1NP were determined at pre-specified time points.
Time Frame: Blood samples were taken Days 1 (baseline), 8, 15, 29, 57, 64, 71, 85, 113, and 169
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
percentage change
  Day 8: number analyzed (Participants) | 4 | 3 | 4 | 5 | 4 | 4
  Day 8 | 19.81 (20.96) | 12.75 (13.03) | 65.12 (17.75) | 31.77 (11.69) | 35.91 (21.89) | 35.35 (47.08)
  Day 15: number analyzed (Participants) | 3 | 4 | 4 | 4 | 4 | 3
  Day 15 | 11.03 (13.94) | 12.43 (13.07) | 52.25 (29.71) | 10.52 (14.72) | 58.58 (54.61) | 28.35 (55.00)
  Day 29: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 29 | 5.24 (12.87) | 6.18 (18.64) | 21.52 (25.01) | 1.96 (9.22) | 32.13 (59.10) | -11.54 (11.35)
  Day 57: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 57 | -2.11 (20.26) | -22.37 (19.82) | 14.57 (36.09) | -6.36 (17.51) | 19.07 (56.24) | -14.26 (12.93)
  Day 64: number analyzed (Participants) | 3 | 4 | 4 | 3 | 3 | 4
  Day 64 | 14.82 (28.86) | 19.12 (40.48) | 39.63 (31.92) | 25.42 (16.73) | 77.17 (109.07) | 17.51 (35.74)
  Day 71: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 4
  Day 71 | 12.19 (21.37) | -5.72 (28.50) | 49.37 (37.99) | 16.79 (12.29) | 42.16 (59.39) | 5.12 (29.54)
  Day 85: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85 | -7.34 (22.50) | -23.50 (13.42) | 26.12 (48.97) | -0.72 (21.29) | 5.79 (23.45) | -11.78 (30.09)
  Day 113: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 113 | -1.13 (13.42) | -13.75 (19.11) | 21.10 (40.61) | 2.53 (42.46) | -5.02 (21.00) | -26.95 (10.23)
  Day 169: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169 | -6.62 (30.96) | -3.13 (10.54) | 18.10 (57.53) | -2.24 (23.99) | -14.30 (19.41) | -21.85 (16.18)

11. Secondary Outcome: Percentage Change From Baseline in Bone Mineral Density (BMD) of the Lumbar Spine
Description: BMD was assessed by dual energy X-ray absorptiometry (DXA) scans of the anteroposterior lumbar spine (L1 through L4) and analyzed by a central imaging laboratory. At least 2 lumbar vertebrae from L1 - L4 must be evaluable by DXA.
Time Frame: DXA scans were during screening (baseline) and at Day 85 and Day 169
Population: The BMD Analysis Set: all participants who have a baseline lumbar spine DXA BMD measurement and at least 1 post-baseline lumbar spine DXA BMD measurement. Participants with data available at each time point are presented.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
percentage change
  Day 85: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85 | 4.84 (3.29) | 7.94 (5.32) | 12.91 (2.60) | 7.78 (9.16) | 7.88 (1.99) | 13.07 (13.45)
  Day 169: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169 | 7.80 (2.23) | 9.24 (7.98) | 15.04 (4.32) | 7.09 (7.03) | 7.10 (6.58) | 12.70 (12.86)

12. Secondary Outcome: Percentage Change From Baseline in Bone Mineral Content (BMC) of the Lumbar Spine
Description: BMC was assessed by DXA scans of the anteroposterior lumbar spine (L1 through L4) and analyzed by a central imaging laboratory. At least 2 lumbar vertebrae from L1 - L4 must be evaluable by DXA.
Time Frame: DXA scans were during screening (baseline) and at Day 85 and Day 169
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
percentage change
  Day 85: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85 | 7.68 (8.10) | 10.13 (6.05) | 18.16 (7.86) | 8.41 (6.90) | 14.62 (3.39) | 16.03 (8.32)
  Day 169: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169 | 12.64 (4.07) | 11.40 (7.82) | 21.29 (11.31) | 7.98 (7.77) | 14.27 (5.52) | 12.42 (10.72)

13. Secondary Outcome: Percentage Change From Baseline in Lumbar Spine Bone Area
Description: Bone area was assessed by DXA scans of the anteroposterior lumbar spine (L1 through L4) and analyzed by a central imaging laboratory. At least 2 lumbar vertebrae from L1 - L4 must be evaluable by DXA.
Time Frame: DXA scans were during screening (baseline) and at Day 85 and Day 169
Population: The BMD Analysis Set: all participants who have a baseline lumbar spine DXA BMD measurement and at least 1 post-baseline lumbar spine DXA BMD measurement.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
percentage change
  Day 85: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 85 | 2.72 (6.99) | 2.03 (1.62) | 4.60 (5.00) | 0.80 (4.62) | 6.23 (2.15) | 3.44 (11.05)
  Day 169: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169 | 4.53 (4.92) | 1.92 (0.66) | 5.30 (6.06) | 0.82 (1.95) | 6.87 (5.14) | -0.09 (4.27)

14. Secondary Outcome: Mean Change From Baseline in Lumbar Spine BMD Z-Score
Description: Lumbar spine BMD was assessed by DXA scans. The results were then converted to Z-scores. The Z-score indicated the number of standard deviations away from the reference population and a score of 0 is equal to the mean. Positive changes from baseline indicated an improvement in lumbar spine BMD.
Time Frame: DXA scans were during screening (baseline) and at Day 85 and Day 169
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 4 | 4
Z-score
  Day 85: number analyzed (Participants) | 4 | 3 | 4 | 4 | 4 | 4
  Day 85 | 0.20 (0.39) | 0.45 (0.37) | 0.50 (0.12) | 0.33 (0.53) | 0.33 (0.26) | 0.53 (0.79)
  Day 169: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4
  Day 169 | 0.33 (0.46) | 0.48 (0.51) | 0.48 (0.21) | 0.25 (0.39) | 0.23 (0.56) | 0.50 (0.62)

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from enrollment to the end of study visit (Day 169); median time on study was 5.55 months. Adverse events were collected from first dose of study drug until the end of study visit (Day 169); median duration was 5.55 months.
Arm/Group | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/5 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 0/4 | 1/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/4 | 2/4 | 4/5 | 1/4 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) (N=4) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) (N=4) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) (N=4) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) (N=5) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) (N=4) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age) (N=4)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Romosozumab Dose A (12 to < 18 Years of Age) (N=4) | Cohort 2: Romosozumab Dose A (5 to < 12 Years of Age) (N=4) | Cohort 3: Romosozumab Dose B (12 to < 18 Years of Age) (N=4) | Cohort 4: Romosozumab Dose B (5 to < 12 Years of Age) (N=5) | Cohort 5: Romosozumab Dose C (12 to < 18 Years of Age) (N=4) | Cohort 6: Romosozumab Dose C (5 to < 12 Years of Age) (N=4)
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT04545554/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT04545554/SAP_001.pdf